CLINICAL TRIAL: NCT00860444
Title: The Heart Healthy and Ethnically Relevant (HHER) Lifestyle Program for Cardiovascular Risk Reduction
Brief Title: Cardiovascular Risk Reduction Program Aimed at African American Women (The HHER Lifestyle Program)
Acronym: HHER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Deborah Parra-Medina, Professor, Epidemiology and Biostatistics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 622; R01HL073001 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Diseases
Keywords: Primary Care; Diet; Physical Activity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will take part in the basic educational and counseling program through their community health care center.
  Interventions: Behavioral: Basic Educational and Counseling Program
- 2 (Experimental): Participants will take part in the comprehensive educational and counseling program through their community health care center.
  Interventions: Behavioral: Comprehensive Educational and Counseling Program

INTERVENTIONS:
Behavioral: Basic Educational and Counseling Program — Participants will receive one session of brief patient-centered physician counseling, along with educational handouts and nurse-assisted guidance with goal-setting.
  Arms: 1
Behavioral: Comprehensive Educational and Counseling Program — Participants will receive one session of brief patient-centered physician counseling, along with educational handouts and nurse-assisted guidance with goal-setting. They will also receive 12 months of telephone counseling and a monthly newsletter.
  Arms: 2

SUMMARY:
Cardiovascular disease (CVD) is a serious health problem among African American women. This study will evaluate a health care center-based program that aims to encourage African American women to eat a low fat diet and increase their physical activity levels to reduce the risk of developing CVD.

DETAILED DESCRIPTION:
CVD is the leading cause of death for women in the United States. It affects African American women at a higher rate than it does white women. People at risk for CVD are encouraged to maintain a healthy weight, eat a healthy diet that is low in fat and cholesterol, and increase their physical activity. Heath care centers are excellent places to provide counseling to people on ways to reduce their risk of CVD. In this study, researchers will evaluate the effectiveness of a community health care center-based counseling program aimed at reducing CVD risk factors among African American women from financially disadvantaged backgrounds.

This study will enroll African American women. Participants will be randomly assigned to one of two groups-either a basic program or a comprehensive program. During a routine, scheduled visit with their health care providers, all participants will learn about the importance of increasing physical activity and eating a low fat diet. All participants will also receive educational materials and a community resource guide. In addition to this, participants in the comprehensive program will receive a pedometer and will be asked to keep a daily log of their physical activity and eating habits. Once a month, these same participants will receive telephone calls from a health counselor and a newsletter by mail that encourages them to maintain a healthy lifestyle. All participants will receive home visits from study staff at baseline and Months 6 and 12. During these visits, participants will undergo blood pressure, weight, height, and waist measurements and a blood collection. Participants will complete questionnaires to assess their medical history, diet, and physical activity habits. For 1 week after each visit, participants will wear a physical activity monitor and keep an activity diary.

ELIGIBILITY:
Inclusion Criteria:

* African American women
* Able and willing to complete survey instruments and assessment procedures

Exclusion Criteria:

* Physical disability or orthopedic problem that limits physical activity
* Elevated blood pressure (i.e., greater than 160/95 mm Hg)
* Insulin-dependent diabetes
* Pregnant or planning to become pregnant during the study period

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Hours per week in moderate and vigorous intensity physical activities (MVPA), as measured by the Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire | Measured at baseline and Months 6 and 12
Weekly consumption frequency of dietary fat and cholesterol, as measured by the New Leaf Dietary Risk Assessment (DRA) | Measured at baseline and Months 6 and 12

SECONDARY OUTCOMES:
Body mass index (weight [kg]/height [m2]) | Measured at baseline and Months 6 and 12
Central adiposity (i.e., waist circumference in inches) | Measured at baseline and Months 6 and 12
Total cholesterol (mg/dL) | Measured at baseline and Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Parra-Medina, PhD, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Background] Parra-Medina D, Wilcox S, Wilson DK, Addy CL, Felton G, Poston MB. Heart Healthy and Ethnically Relevant (HHER) Lifestyle trial for improving diet and physical activity in underserved African American women. Contemp Clin Trials. 2010 Jan;31(1):92-104. doi: 10.1016/j.cct.2009.09.006. Epub 2009 Sep 22. PMID 19781665
- [Result] Parra-Medina D, Wilcox S, Salinas J, Addy C, Fore E, Poston M, Wilson DK. Results of the Heart Healthy and Ethnically Relevant Lifestyle trial: a cardiovascular risk reduction intervention for African American women attending community health centers. Am J Public Health. 2011 Oct;101(10):1914-21. doi: 10.2105/AJPH.2011.300151. Epub 2011 Aug 18. PMID 21852629
- [Result] Wilcox S, Parra-Medina D, Felton GM, Poston MB, McClain A. Adoption and implementation of physical activity and dietary counseling by community health center providers and nurses. J Phys Act Health. 2010 Sep;7(5):602-12. doi: 10.1123/jpah.7.5.602. PMID 20864755